CLINICAL TRIAL: NCT01359943
Title: A Randomized, Double-blind, Placebo-controlled Study of Efficacy, Safety and Tolerability of Secukinumab at 12 Weeks Administered With an Intravenous (i.v.) or Subcutaneous (s.c.) Loading Regimen Compared to Placebo in Patients With Active Rheumatoid Arthritis Despite Treatment With Methotrexate
Brief Title: Efficacy, Safety and Tolerability of Secukinumab in Patients With Rheumatoid Arthritis Taking Methotrexate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAIN457F2206; 2010-024516-34 (EudraCT Number)
Record Dates: First submitted 2011-05-19; First posted 2011-05-25 (Estimated); Results first posted 2015-03-02 (Estimated); Last update posted 2015-03-02 (Estimated); Status verified 2015-02

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; RA; secukinumab; AIN457; inflammatory joints; American College of Rheumatology; ACR
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — secukinumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- secukinumab 10 mg/kg i.v. loading (Experimental): secukinumab 10mg/kg i.v. loading at Weeks 0, 2 and 4, and placebo s.c. at weeks 0, 1, 2, 3 and 4, followed by secukinumab 150mg s.c. every 4 weeks starting at Week 8
  Interventions: Biological: secukinumab (AIN457); Drug: placebo
- secukinumab 150 mg s.c. loading (Experimental): secukinumab 150mg s.c. loading at Weeks 0, 1, 2, 3 and 4, and placebo i.v. at weeks 0, 2 and 4, followed by secukinumab 150mg s.c. every 4 weeks starting at Week 8
  Interventions: Biological: secukinumab (AIN457); Drug: placebo
- placebo (Placebo Comparator): placebo at Weeks 0, 1, 2, 3, 4, 8 & 12, followed by secukinumab 150mg s.c. every 4 weeks starting at Week 16
  Interventions: Biological: secukinumab (AIN457); Drug: placebo

INTERVENTIONS:
Biological: secukinumab (AIN457) — Secukinumab is a human monoclonal antibody. Monoclonal antibodies are proteins that recognize and bind to unique proteins that your body produces. Secukinumab binds and reduces the activity of a cytokine (a "messenger" protein in the body) called Interleukin 17 (IL-17).
Drug: placebo — Matching placebo to AIN457 i.v. and to AIN457 s.c..

SUMMARY:
The study compared the efficacy and assessed the safety of secukinumab given as 3 intravenous (i.v.) loading doses or weekly sub-cutaneous (s.c.) loading doses, compared to placebo, followed by monthly s.c. injections in patients with active Rheumatoid Arthritis (RA) despite treatment with Methotrexate.

ELIGIBILITY:
Inclusion criteria:

* presence of RA classified by ACR 2010 revised criteria for at least 3 months before screening
* must have been taking MTX for at least 3 months before randomization and must currently be on a stable dose of MTX for at least 4 weeks before randomization.
* At Baseline: Disease activity criteria defined by >6 tender joints out of 68 and >6 swollen joints out of 66 and with at least 1 of the following at screening: Anti-CCP antibodies positive OR Rheumatoid Factor positive and with at least 1 of the following at screening: hsCRP ≥ 10 mg/L OR ESR ≥ 28

Exclusion criteria:

* RA patients functional status class IV according to the ACR 1991 revised criteria
* Previous exposure to secukinumab or any other biologic drug directly targeting IL-17 or IL-17 receptor
* Previous exposure ever to an anti-TNF-a agent or any other immunomodulatory biologic agent (experimental or approved)
* Patients taking high potency opioid analgesics (e.g., methadone, hydromorphone, or morphine)
* Any therapy by intra-articular injections (e.g. corticosteroid, hyaluronan) required for treatment of arthritis within 4 weeks before randomization
* Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2011-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals; Novartis Pharmceuticals, Study Director — Novartis Pharmaceuticals
Locations (35):
- United States (8):
  - Novartis Investigative Site, Vestavia Hills, Alabama
  - Novartis Investigative Site, Peoria, Arizona
  - Novartis Investigative Site, Upland, California
  - Novartis Investigative Site, Bowling Green, Kentucky
  - Novartis Investigative Site, Tupelo, Mississippi
  - Novartis Investigative Site, Lincoln, Nebraska
  - Novartis Investigative Site, Jackson, Tennessee
  - Novartis Investigative Site, Nashville, Tennessee
- Bulgaria (4):
  - Novartis Investigative Site, Pleven, Bulgaria
  - Novartis Investigative Site, Plovdiv, Bulgaria
  - Novartis Investigative Site, Sevlievo, Bulgaria
  - Novartis Investigative Site, Sofia, Bulgaria
- Canada (2):
  - Novartis Investigative Site, St. John's, Newfoundland and Labrador
  - Novartis Investigative Site, Sainte-Foy, Quebec
- Hungary (3):
  - Novartis Investigative Site, Szeged, Hungary
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
- Italy (6):
  - Novartis Investigative Site, Valeggio sul Mincio, (vr)
  - Novartis Investigative Site, Arenzano, GE
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Siena, SI
  - Novartis Investigative Site, Torino, TO
- Poland (3):
  - Novartis Investigative Site, Bialystok
  - Novartis Investigative Site, Poznan
  - Novartis Investigative Site, Warsaw
- Novartis Investigative Site, San Juan, Puerto Rico
- Slovakia (8):
  - Novartis Investigative Site, Bardejov, Slovak Republic
  - Novartis Investigative Site, Lučenec, Slovakia
  - Novartis Investigative Site, Partizánske, Slovakia
  - Novartis Investigative Site, Piešťany, Slovakia
  - Novartis Investigative Site, Sabinov, Slovakia
  - Novartis Investigative Site, Stará Ľubovňa, Slovakia
  - Novartis Investigative Site, Topoľčany, Slovakia
  - Novartis Investigative Site, Trnava, Slovensko

REFERENCES:
- [Derived] Tlustochowicz W, Rahman P, Seriolo B, Krammer G, Porter B, Widmer A, Richards HB. Efficacy and Safety of Subcutaneous and Intravenous Loading Dose Regimens of Secukinumab in Patients with Active Rheumatoid Arthritis: Results from a Randomized Phase II Study. J Rheumatol. 2016 Mar;43(3):495-503. doi: 10.3899/jrheum.150117. Epub 2016 Feb 1. PMID 26834211

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were randomized to one of the following 3 treatment groups in a 2:2:1 ratio: secukinumab 10 mg/kg i.v., secukinumab 150 mg s.c. or placebo.
Period: Double-blind (Weeks 0 - 16)
Arm/Group | Secukinumab 10 mg/kg i.v. Loading | Secukinumab 150 mg s.c. Loading | Placebo
Started | 88 | 89 | 44
Completed | 86 | 85 | 44
Not Completed | 2 | 4 | 0
Not completed — Abnormal laboratory values | 1 | 0 | 0
Not completed — Adverse Event | 1 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 0
Period: Open Label 150 mg s.c. (Weeks 16 - 52)
Arm/Group | Secukinumab 10 mg/kg i.v. Loading | Secukinumab 150 mg s.c. Loading | Placebo
Started | 86 | 84 (One participant, who was continuing as of week 12, did not receive study drug at week 16.) | 44
Completed | 78 | 71 | 36
Not Completed | 8 | 13 | 8
Not completed — Administrative problems | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 3 | 4
Not completed — Protocol deviation | 0 | 1 | 0
Not completed — Lack of Efficacy | 3 | 3 | 3
Not completed — Abnormal laboratory values | 0 | 1 | 0
Not completed — Adverse Event | 3 | 5 | 1
Period: Follow-up (Weeks 52 - 60)
Arm/Group | Secukinumab 10 mg/kg i.v. Loading | Secukinumab 150 mg s.c. Loading | Placebo
Started | 86 | 84 | 44
Completed | 78 | 69 | 36
Not Completed | 8 | 15 | 8
Not completed — Withdrawal by Subject | 1 | 5 | 4
Not completed — Administrative problems | 1 | 0 | 0
Not completed — Protocol deviation | 0 | 1 | 0
Not completed — Lack of Efficacy | 3 | 3 | 3
Not completed — Abnormal laboratory value | 0 | 1 | 0
Not completed — Adverse Event | 3 | 5 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Secukinumab 10 mg/kg i.v. Loading | Secukinumab 150 mg s.c. Loading | Placebo | Total
Number analyzed (Participants) | 88 | 89 | 44 | 221
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.8 (11.81) | 54.5 (12.26) | 53.5 (9.33) | 54.0 (11.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 72 | 37 | 176
  Male | 21 | 17 | 7 | 45

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieve American College of Rheumatology Response of 20 (ACR20)
Description: A participant was considered to be a responder according to the ACR20 criteria if the participant had at least 20% improvement in both the tender joint count and swollen joint count measures, and in at least 3 of the following 5 measures: patient's assessment of pain, patient's global assessment of disease activity, physician's global assessment of disease activity, Health Assessment Questionnaire (HAQ©) score, and/or C-reactive protein (CRP)/Erythrocyte Sedimentation Rate (ESR).
Time Frame: 12 weeks
Population: Full analysis set (FAS): The FAS included all participants who were randomized to study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Secukinumab 10 mg/kg i.v. Loading | Secukinumab 150 mg s.c. Loading | Placebo
Number analyzed (Participants) | 88 | 89 | 44
Percentage of participants | 53.4 | 44.9 | 40.9

2. Secondary Outcome: Percentage of Participants Who Achieve ACR50 and ACR70
Description: A participant was considered to be a responder according to the ACR50 or ACR70 criteria if the participant had at least 50% or 70% improvement, respectively, in both the tender joint count and swollen joint count measures, and in at least 3 of the following 5 measures: patient's assessment of pain, patient's global assessment of disease activity, physician's global assessment of disease activity, Health Assessment Questionnaire (HAQ©) score, and/or C-reactive protein (CRP)/Erythrocyte Sedimentation Rate (ESR).
Time Frame: 12 weeks
Population: Full analysis set (FAS): The FAS included all participants who were randomized to study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Secukinumab 10 mg/kg i.v. Loading | Secukinumab 150 mg s.c. Loading | Placebo
Number analyzed (Participants) | 88 | 89 | 44
Percentage of participants
  ACR50 | 20.5 | 18.0 | 11.4
  ACR70 | 8.0 | 5.6 | 0.0

3. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire-Disease Index (HAQ-DI) Score.
Description: The HAQ measures physical disability and functional status. It has 4 dimensions: disability, pain, drug side effects and dollar costs. In this trial, only the disability dimension was used. The disability dimension consists of 20 multiple choice items concerning difficulty in performing 8 common activities of daily living; dressing and grooming, arising, eating, walking, reaching, personal hygiene, gripping and activities. Participants choose from four response categories: 0 (without any difficulty), 1 (with some difficulty), 2 (with much difficulty) and 3 (unable to do). Within each of the 8 categories, only the item indicating the most severe impairment contributes to the category score. The HAQ score is calculated by summing the computed scores for each category and dividing by the number of categories answered. It ranges from 0 (without any difficulty) to 3 (unable to do). A negative change from baseline indicates improvement.
Time Frame: baseline, 12 Weeks
Population: Full analysis set (FAS): The FAS included all participants who were randomized to study treatment.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Secukinumab 10 mg/kg i.v. Loading | Secukinumab 150 mg s.c. Loading | Placebo
Number analyzed (Participants) | 88 | 89 | 44
score on a scale | -0.35 (0.052) | -0.28 (0.053) | -0.17 (0.074)

4. Secondary Outcome: Change From Baseline in DAS28 Using High Sensitivity C-reactive Protein (hsCRP) (DAS28-CRP)
Description: The Disease Activity Score (DAS) is a combined index to measure disease activity in RA participants. DAS28-CRP is determined using the following variables: 28-joint counts (tender28 and swollen28), CRP, and the participant's general health (GH) or global disease activity measured on a Visual Analogue Scale (VAS) of 100 mm (0 = and 100 = ). Using the data from these variables, DAS28-CRP is calculated using the following formula: DAS28-4(crp) = 0.56*sqrt(TJC28) + 0.28*sqrt(SJC28) + 0.36*ln(CRP+1) + 0.014*GH + 0.96. The calculation results in a DAS28-CRP score from 0 to 10 indicating the current activity of the rheumatoid arthritis of your patient. A DAS28 above 5.1 means high disease activity whereas a DAS28 below 3.2 indicates low disease activity. Remission is achieved by a DAS28 lower than 2.6. A negative change from baseline indicates improvement.
Time Frame: baseline, 12 weeks
Population: Participants from the full analysis set (FAS), who had values at both baseline and week 12, were included in this analysis. The FAS included all participants who were randomized to study treatment.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Secukinumab 10 mg/kg i.v. Loading | Secukinumab 150 mg s.c. Loading | Placebo
Number analyzed (Participants) | 85 | 82 | 43
score on a scale | -1.67 (0.119) | -1.65 (0.120) | -1.21 (0.166)

5. Secondary Outcome: Change From Baseline in Disease Activity Score 28 Response Using ESR (DAS28-ESR)
Description: The Disease Activity Score (DAS) is a combined index to measure disease activity in RA participants. DAS28 is determined using the following variables: 28-joint counts (tender28 and swollen28), erythrocyte sedimentation rate (ESR), and the participant's general health (GH) or global disease activity measured on a Visual Analogue Scale (VAS) of 100 mm (0 = and 100 = ). Using the data from these variables, DAS28-ESR is calculated using the following formula: DAS28 = 0.56 * sqrt(tender28) + 0.28 * sqrt(swollen28) + 0.70 * ln(ESR) + 0.014 * GH. The calculation results in a DAS28-ESR score from 0 to 10 indicating the current activity of the rheumatoid arthritis of your patient. A DAS28 above 5.1 means high disease activity whereas a DAS28 below 3.2 indicates low disease activity. Remission is achieved by a DAS28 lower than 2.6. A negative change from baseline indicates improvement.
Time Frame: baseline, 12 weeks
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Secukinumab 10 mg/kg i.v. Loading | Secukinumab 150 mg s.c. Loading | Placebo
Number analyzed (Participants) | 84 | 82 | 43
score on a scale | -1.98 (0.126) | -1.80 (0.128) | -1.46 (0.179)

6. Secondary Outcome: Percentage of Participants With European League Against Rheumatism (EULAR) Response
Description: EULAR response criteria are based on DAS28 status in combination with DAS28 improvements. The EULAR response criteria are as follows: present DAS28 <3.2 with DAS28 improvement >1.2 corresponds to 'good response'; present DAS28 <3.2 with DAS28 improvement between 0.6 to 1.2, or present DAS28 between 3.2 to 5.1 with DAS28 improvement from 0.6 to >1.2, or present DAS28 >5.2 with DAS28 improvement >1.2 correspond to 'moderate response; present DAS28 <3.2 with DAS28 improvement <0.6, or present DAS28 between 3.2 to 5.1 with DAS28 improvement <0.6, or present DAS28 >5.1 with DAS28 improvement <0.6 to 1.2 correspond to 'no response'.
Time Frame: baseline, 12 weeks
Population: Full analysis set (FAS): The FAS included all participants who were randomized to study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Secukinumab 10 mg/kg i.v. Loading | Secukinumab 150 mg s.c. Loading | Placebo
Number analyzed (Participants) | 88 | 89 | 44
Percentage of participants
  Good response | 28.4 | 27.0 | 13.6
  Moderate response | 46.6 | 44.9 | 52.3
  No response | 25.0 | 28.1 | 34.1

7. Secondary Outcome: Change From Baseline in Swollen 66-joint Count
Description: The 66 joints assessed for swelling included the 8 distal interphalangeal, 10 proximal interphalangeal and 10 metacarpophalangeal joints of the hands, the 10 metatarsophalangeal and 10 proximal interphalangeal joints of the feet, the 2 wrists, 2 elbows , 2 shoulders , 2 acromioclavicular, 2 sternoclavicular, 2 temporomandibular, 2 knee, 2 talo-tibial, and 2 mid-tarsal joints. Swelling was graded present (1) or absent (0). A negative change in baseline indicates improvement.
Time Frame: baseline, 12 weeks
Population: Full analysis set (FAS): The FAS included all participants who were randomized to study treatment.
Measure: Least Squares Mean (Standard Error); unit: Number of joints
Arm/Group | Secukinumab 10 mg/kg i.v. Loading | Secukinumab 150 mg s.c. Loading | Placebo
Number analyzed (Participants) | 88 | 89 | 44
Number of joints | -9.49 (0.607) | -9.81 (0.612) | -7.88 (0.863)

8. Secondary Outcome: Change From Baseline in Tender 68-joint Count
Description: The 68 joints assessed for tenderness included the 8 distal interphalangeal, 10 proximal interphalangeal and 10 metacarpophalangeal joints of the hands, the 10 metatarsophalangeal and 10 proximal interphalangeal joints of the feet, the 2 wrists, 2 elbows , 2 shoulders , 2 acromioclavicular, 2 sternoclavicular, 2 temporomandibular, 2 hip, 2 knee, 2 talo-tibial, and 2 mid-tarsal joints. Joint tenderness was graded present (1) or absent (0). A negative change from baseline indicates improvement.
Time Frame: baseline, 12 weeks
Population: Full analysis set (FAS): The FAS included all participants who were randomized to study treatment.
Measure: Least Squares Mean (Standard Error); unit: Number of joints
Arm/Group | Secukinumab 10 mg/kg i.v. Loading | Secukinumab 150 mg s.c. Loading | Placebo
Number analyzed (Participants) | 88 | 89 | 44
Number of joints | -10.31 (1.093) | -11.99 (1.099) | -9.50 (1.549)

9. Secondary Outcome: Change From Baseline in Participant's Assessment of Rheumatoid Arthritis (RA) Pain
Description: The patient's assessment of pain was performed using 100 mm visual analog scale (VAS) ranging from 0 (no pain) to 100 (unbearable pain) after the question "Please indicate with a vertical mark through the horizontal line the most pain you had from your rheumatoid arthritis over the last 24 hours". A negative change from baseline indicates improvement.
Time Frame: baseline, 12 weeks
Population: Full analysis set (FAS): The FAS included all participants who were randomized to study treatment.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Secukinumab 10 mg/kg i.v. Loading | Secukinumab 150 mg s.c. Loading | Placebo
Number analyzed (Participants) | 88 | 89 | 44
score on a scale | -14.41 (2.057) | -12.60 (2.071) | -6.66 (2.902)

10. Secondary Outcome: Change From Baseline in Participant's Global Assessment of Disease Activity
Description: The patient's global assessment of disease activity was performed using 100 mm VAS ranging from 0 (very good) to 100 (very poor), after the question "Considering all the ways rheumatoid arthritis affects you, please indicate with a vertical mark through the horizontal line how well you are doing today". A negative change from baseline indicates improvement.
Time Frame: baseline, 12 weeks
Population: Full analysis set (FAS): The FAS included all participants who were randomized to study treatment.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Secukinumab 10 mg/kg i.v. Loading | Secukinumab 150 mg s.c. Loading | Placebo
Number analyzed (Participants) | 88 | 89 | 44
score on a scale | -18.58 (2.042) | -15.29 (2.063) | -9.93 (2.884)

11. Secondary Outcome: Change From Baseline in Physician's Global Assessment of Disease Activity
Description: The physician's global assessment of disease activity was performed using 100 mm VAS ranging from 0 (very good) to 100 (very poor), after the question "Considering all the ways rheumatoid arthritis affects your patient, how would you rate his or her current condition?". A negative change from baseline indicates improvement.
Time Frame: baseline, 12 weeks
Population: Full analysis set (FAS): The FAS included all participants who were randomized to study treatment.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Secukinumab 10 mg/kg i.v. Loading | Secukinumab 150 mg s.c. Loading | Placebo
Number analyzed (Participants) | 88 | 89 | 44
score on a scale | -27.05 (1.925) | -29.01 (1.950) | 18.88 (2.726)

12. Secondary Outcome: Change From Baseline in hsCRP
Description: Blood for this assessment was obtained to identify the presence of inflammation, to determine its severity, and to monitor response to treatment. A negative change from baseline indicates improvement.
Time Frame: baseline, 12 weeks
Population: Full analysis set (FAS): The FAS included all participants who were randomized to study treatment.
Measure: Least Squares Mean (Standard Error); unit: mg/L
Arm/Group | Secukinumab 10 mg/kg i.v. Loading | Secukinumab 150 mg s.c. Loading | Placebo
Number analyzed (Participants) | 88 | 89 | 44
mg/L | -6.00 (0.938) | -5.72 (0.946) | -1.69 (1.336)

13. Secondary Outcome: Change From Baseline in ESR
Description: Blood for this assessment was obtained to monitor disease activity and response to therapy. A negative change from baseline indicates improvement.
Time Frame: baseline, 12 weeks
Population: Full analysis set (FAS): The FAS included all participants who were randomized to study treatment.
Measure: Least Squares Mean (Standard Error); unit: mm/hr
Arm/Group | Secukinumab 10 mg/kg i.v. Loading | Secukinumab 150 mg s.c. Loading | Placebo
Number analyzed (Participants) | 88 | 89 | 44
mm/hr | -16.68 (1.409) | -12.43 (1.425) | -10.53 (1.993)

ADVERSE EVENTS:
Groups:
- AIN457 Pooled Treatment Groups - Open Label Period: Week 16 through week 52: AIN457 150 mg s.c. open label
- AIN457 Pooled Treatment Groups - Follow-up Period: Follow-up period: week 52 through week 60 - AIN457 150 mg sc open label
Arm/Group | Secukinumab 10 mg/kg i.v. Loading | Secukinumab 150 mg s.c. Loading | Placebo | AIN457 Pooled Treatment Groups - Open Label Period | AIN457 Pooled Treatment Groups - Follow-up Period
Serious Adverse Events (participants affected / at risk) | 2/88 | 3/89 | 1/44 | 18/214 | 3/214
Other Adverse Events (participants affected / at risk) | 17/88 | 30/89 | 18/44 | 78/214 | 10/214
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Secukinumab 10 mg/kg i.v. Loading (N=88) | Secukinumab 150 mg s.c. Loading (N=89) | Placebo (N=44) | AIN457 Pooled Treatment Groups - Open Label Period (N=214) | AIN457 Pooled Treatment Groups - Follow-up Period (N=214)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Arteriogram coronary (Investigations) | 0 | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Lumbar radiculopathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Rheumatoid lung (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Secukinumab 10 mg/kg i.v. Loading (N=88) | Secukinumab 150 mg s.c. Loading (N=89) | Placebo (N=44) | AIN457 Pooled Treatment Groups - Open Label Period (N=214) | AIN457 Pooled Treatment Groups - Follow-up Period (N=214)
Leukopenia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0 | 5 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 1 | 0 | 2 | 0
Immunodeficiency (Immune system disorders) | 0 | 0 | 1 | 0 | 0
Cystitis (Infections and infestations) | 0 | 2 | 0 | 2 | 0
Erythema migrans (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 2 | 1 | 1 | 3 | 0
Influenza (Infections and infestations) | 0 | 1 | 1 | 4 | 0
Laryngitis (Infections and infestations) | 1 | 2 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 5 | 5 | 4 | 11 | 1
Oral herpes (Infections and infestations) | 0 | 1 | 3 | 5 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 6 | 1
Rhinitis (Infections and infestations) | 2 | 0 | 2 | 3 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 17 | 1
Urinary tract infection (Infections and infestations) | 0 | 2 | 1 | 3 | 0
Haemoglobin decreased (Investigations) | 0 | 1 | 1 | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 2 | 0 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1 | 2
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 5 | 2 | 12 | 5
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 5 | 0
Headache (Nervous system disorders) | 2 | 4 | 1 | 5 | 0
Sciatica (Nervous system disorders) | 2 | 0 | 0 | 2 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Mood altered (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 1 | 3 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 7 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 3 | 0
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 2 | 1 | 11 | 0
Varicose vein (Vascular disorders) | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.